CLINICAL TRIAL: NCT06723158
Title: Investigating the Impact of Virtual Reality Glasses on Sedation Requirement and Patient Experience in Patients Undergoing Oral Surgery
Brief Title: Oral Surgery Virtual Reality Glasses Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-45038
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Procedural Anxiety; Procedural Pain
Keywords: Virtual reality glasses; Non emergent oral surgery; IV sedation; Patient Health Questionnaire (PHQ); Generalized Anxiety Disorder (GAD)
MeSH Terms: conditions — Pain, Procedural; Generalized Anxiety Disorder | interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: Randomized group allocation (1:1 block size of 2 for randomization)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) Intervention Group (Experimental): Participants randomized to this group will receive VR glasses with a relaxation module (audio, visual) to wear during IV placement, induction of anesthesia, and during the procedure.
  Interventions: Other: Virtual reality (VR) glasses with relaxation module
- Virtual Reality (VR) Control Group (No Intervention): Participants randomized to this group will receive VR glasses without a relaxation module to be worn only as safety glasses, during IV placement, induction of anesthesia, and during the procedure.

INTERVENTIONS:
Other: Virtual reality (VR) glasses with relaxation module — The relaxation module will include immersive video and audio components as a distraction from the medical procedures.
  Arms: Virtual Reality (VR) Intervention Group

SUMMARY:
The goal of this randomized trial is to investigate if using virtual reality (VR) glasses for patients who require non-emergent oral surgery procedures under intravenous (IV) sedation improves their overall experience compared to using standard of care safety glasses.

This study has two primary objectives.

1. To evaluate if VR glasses can improve patient tolerance during IV access, sedation induction, and the surgical procedure.
2. To investigate whether the use of VR glasses reduces the amount of sedation required for induction and throughout the oral surgery procedure.

80 subjects will be randomly assigned 1:1 to either wear VR glasses playing a relaxing video and audio or VR glasses that will only serve as eye protection (control group).

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring IV sedation for oral surgery procedure
* Patients able to understand the use of virtual reality glasses and provide informed consent/assent
* Patients classified as American Society of Anesthesiologists (ASA) I or II
* No reported substance use within the previous 24 hours
* No reported excessive alcohol consumption
* Willingness to wear eye protection
* Willingness to use certified interpreters if required
* A legal guardian must accompany minors

Exclusion Criteria:

* Patient with hearing aids or severe hearing impairment
* Patient with blindness or significant visual impairment that is not corrected by contact lenses
* Patients with cognitive impairments determined and assessed by the researchers
* Pregnant women or women who could be pregnant based on self reporting
* Patients unable to tolerate virtual reality glasses due to motion sickness or other issues
* Patients with history of seizures or epilepsy per self report
* Patients who cannot tolerate VR glasses due to discomfort or a medical emergency that arises during the procedure

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-11-18 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Level of anxiety | 3 days before oral surgery, immediately before surgery, immediately after surgery, about 8 hours after surgery
  Scores from the General Anxiety Disorder-7 (GAD-7) will be used to assess the level of anxiety. It is a 7-item instrument with each item scored from 0=Not at all to 3=Nearly every day. GAD-7 total scores for the can range from 0 to 21 with higher scores suggesting more anxiety. The scores are interpreted as 0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, and 15-21: severe anxiety.
Level of depression | 3 days before oral surgery, immediately before surgery, immediately after surgery, about 8 hours after surgery
  Scores from the Patient Health Questionnaire (PHQ-9) will be used to assess the level of depression. It is a 9-item depression screening tool with each item scored from 0=Not at all to 3=Nearly every day. Scores can range from 0 to 27, with higher scores suggesting more depression. The scores are interpreted as 0-4: None or minimal depression, 5-9: Mild depression, 10-14: Moderate depression, 15-19: Moderately severe depression, and 20-27: Severe depression.
Amount of Midazolam used | pre-incision, 30 minutes post incision, 60 minutes post incision
  The amount of this drug used will be abstracted form the medical record of each participant.
Amount of Fentanyl used | pre-incision, 30 minutes post incision, 60 minutes post incision
  The amount of this drug used will be abstracted form the medical record of each participant.
Amount of Propofol used | pre-incision, 30 minutes post incision, 60 minutes post incision
  The amount of this drug used will be abstracted form the medical record of each participant.
Amount of Ketamine used | pre-incision, 30 minutes post incision, 60 minutes post incision
  The amount of this drug used will be abstracted form the medical record of each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Radhika Chigurupati, DMD MS, Principal Investigator — Goldman School of Dental Medicine, Oral and Maxillofacial Surgery
Locations (1):
- Goldman School of Dental Medicine, Oral and Maxillofacial Surgery Clinic, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No